CLINICAL TRIAL: NCT06461156
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HS-10504 in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC）
Brief Title: A Study of HS-10504 in Patients With Advanced or Metastatic Non-Small-Cell Lung Cancer(NSCLC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10504-101
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Metastatic NSCLC
Keywords: locally advanced or metastatic NSCLC; EGFR C797S; HS-10504
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10504 (Experimental): Subjects with advanced or metastatic NSCLC will be enrolled in dose-escalation stage. Dose escalation of HS-10504 will be done to determine maximum tolerated dose(Dose Escalation Stage).
  Depending on data obtained from the dose-escalation stage, dose expansion may proceed with in subjects with advanced or metastatic NSCLC having an EGFR C797S mutation. It can be conducted at the potentially safe and effective doses(Dose Expansion Stage).
  Interventions: Drug: HS-10504

INTERVENTIONS:
Drug: HS-10504 — HS-10504 will be administered orally once daily in a continuous regimen. Participants will continue treatment until experiencing objective disease progression or meeting other protocol-specified criteria for discontinuation of study treatment.

SUMMARY:
HS-10504 is a fourth-generation epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor targeting EGFR C797S mutation. This study will evaluate the safety, tolerability, pharmacokinetics and efficacy of HS-10504 in Chinese locally advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged ≥ 18 years.
* Subjects with histologically or cytologically confirmed locally advanced or metastatic NSCLC
* Progressive disease on or after prior treatment with EGFR-TKIs.
* Enrollment will be restricted to participants with evidence of EGFR-positive in tumor as determined by local or central testing.
* At least 1 target lesion according to RECIST 1.1.
* ECOG PS score: 0-1.
* Estimated life expectancy> 12 weeks.
* Men or women should be using adequate contraceptive measures throughout the study.
* Women must have the evidence of non-childbearing potential.
* Signed and dated Informed Consent Form.

Exclusion Criteria:

* Subjects with known oncogenic driver genes other than EGFR.
* Subjects with mixed cell histologic or with phenotypic transformation.
* Treatment with any of the following:

  1. Prior or concurrent treatment with fourth-generation EGFR tyrosine kinase inhibitors.
  2. Cytotoxic chemotherapy, any other investigational drugs, traditional Chinese medicine with anti-tumor indications, or other anti-tumor drugs within 14 days prior to the first dose of HS-10504 or require continued treatment with these drugs during the study.
  3. Any local radiotherapy 2 weeks prior to the first dose of study treatment; have received irradiation of more than 30% of bone marrow prior to the first dose
  4. Uncontrolled pleural effusion or ascites or pericardial effusion.
  5. Major surgery within 4 weeks before the first dose.
  6. CNS metastases with symptomatic or active progression.
* Subjects who have any grade ≥2 residual toxicities from prior therapies.
* Subjects who have history of other primary malignancies.
* Inadequate bone marrow reserve or hepatic and renal functions.
* Subjects with severe or poorly controlled diabetes, cardiovascular diseases or hypertension; subjects with severe arteriovenous thrombotic events, severe infection, clinically significant bleeding symptoms or clinically significant gastrointestinal dysfunction.
* Hypersensitivity to any ingredient of HS-10504.
* Moderate to severe pulmonary diseases.
* Prior history of significant neurological or mental disorders.
* Women who are breastfeeding or pregnant or planned to be pregnant during the study period.
* Unlikely to comply with study procedures, restrictions, and requirements in the opinion of the investigator.
* Any disease or condition that, in the opinion of the investigator, would compromise subject safety or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
the maximum tolerated dose (MTD) or the maximum applicable dose (MAD) | From the single dose to the last dose of the first cycle defined as 21 days of multiple dosing (21 days).
  To determine the MTD or MAD for further evaluation of oral administration of HS-10504 in subjects with NSCLC

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs). | From the first dose until 28 days after the last dose
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, and NCI CTCAE v5.0.
maximum plasma concentration (Cmax) of HS-10504 (and its major matabolite) for the first dose and multiple dose adminitration of HS-10504 | From the first dose until Circle 2 Day 1
  Cmax is the maximum observed concentration
Time to reach maximum plasma concentration (Tmax) for the first dose and multiple adminitration of HS-10504 (and its major matabolite) | From the first dose until Circle 2 Day 1
  Tmax is defined as time to reach maximum observed plasma concentration
half-life (T1/2) of HS-10504 (and its major matabolite) for the first dose and multiple dose adminitration of HS-10504 | From the first dose until Circle 2 Day 1
  half-life is the time measured for the concentration to decrease by one half
Area under the curve (AUC) of HS-10504 (and its major matabolite) for the first dose and multiple dose adminitration of HS-10504 | From the first dose until Circle 2 Day 1
  The AUC is defined as the area under the plasma concentration-time curve
Trough plasma concentration (Ctrough) of HS-10504 (and its major matabolite) | From the first dose to disease progression or withdrawal from study, whichever came first, assessed up to 24 months
  Ctrough is the observed plasma concentration immediately prior to the next dose administration
Objective response rate (ORR) | up to 24 months
  ORR was defined as the percentage of participants who achieved a best overall response (BOR) of confirmed Complete Response (CR) or Partial Response (PR), assessed by investigators based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Disease Control Rate (DCR) | up to 24 months
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline. DCR was evaluated by the number of participants with best overall response of CR, PR and stable disease (SD)
Duration of response (DOR) | up to 24 months
  Duration of response (DoR) determined by investigators according to RECIST 1.1. DoR was defined as the period from the first occurrence of CR or PR to progressive disease (PD) or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used
Progression-free survival (PFS) | From the first dose to disease progression or withdrawal from study, whichever came first, assessed up to 24 months
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate progression free survival. Progression-free survival was deﬁned as the time from date of ﬁrst dose until the documentation of objective PD or death from any cause in the absence of progression (whichever occurred first), regardless of whether they subsequently received non-study anti-cancer therapy.
Overall survival (OS), only for dose-expansion stage subjects | From the first dose up to death or withdrawal from study, whichever came first, assessed up to 24 months
  OS was defined as the time from the first dose or random assignment (if any) to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No